CLINICAL TRIAL: NCT06861361
Title: Surgical Bioprosthesis Aortic Valve Replacement Vs. Myval Balloon-Expandable THV Series in Patients Aged 65 to 75 With Symptomatic Severe Aortic Stenosis Judged Eligible by Heart Team
Brief Title: Surgical vs Transcatheter Aortic Valve Replacement in Young Patients
Acronym: START YOUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: START YOUNG
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Severe Aortic Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVR: Myval balloon-expandable THV Series (Experimental): Myval balloon-expandable THV Series will be used for valve replacement
  Interventions: Device: Myval balloon-expandable THV Series
- SAVR: Any surgical bioprosthetic valve commercially available at the clinical investigation site (Active Comparator): Surgical bioprosthetic valve commercially available at the clinical investigation site will be used for valve replacement
  Interventions: Device: Surgical bioprosthetic valve

INTERVENTIONS:
Device: Myval balloon-expandable THV Series — Patients receive Myval balloon-expandable THV Series (TAVR)
  Arms: TAVR: Myval balloon-expandable THV Series
Device: Surgical bioprosthetic valve — Patients receive any surgical bioprosthetic valve commercially available at the clinical investigation site (SAVR)
  Arms: SAVR: Any surgical bioprosthetic valve commercially available at the clinical investigation site

SUMMARY:
The study objective is to demonstrate that the clinical outcomes of the Myval balloon-expandable THV series are non-inferior to those of SAVR in patients with symptomatic severe aortic stenosis aged 65 to 75 years.

DETAILED DESCRIPTION:
Prospective, randomized, multinational, multicenter, open label, trial of 1180 patients treated with surgical bioprosthetic aortic valve replacement (SAVR) or transcatheter aortic valve replacement (TAVR).

ELIGIBILITY:
Inclusion Criteria:

Participant will be included if all the following criteria are met:

1. Patients aged ≥65 and ≤75
2. Symptomatic severe aortic stenosis (mean gradient≥40mmHg, and or peak velocity>4m/sec).
3. Patients with symptomatic heart disease due to severe native calcific aortic stenosis, as judged by a multidisciplinary heart team (including a cardiac surgeon), for whom SAVR or transfemoral TAVR is deemed feasible and approved by the local heart team.Signed informed consent for participation in the clinical investigation

Exclusion Criteria:

Participant will not be included if any one of the following conditions exists:

1. Unable to understand and follow clinical investigation-related instructions or unable to comply with the clinical investigation protocol
2. Life expectancy less than 1 year
3. Known hypersensitivity or allergy to aspirin, clopidogrel or any Device frame components.
4. Under judicial protection, tutorship, or curatorship
5. Participation in another trial before the primary endpoint

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1180 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint at 1 month (non-inferiority): Composite measure of all-cause death, any stroke, bleeding, AKI stage 2-4, rehospitalization for a procedure-related event or or reintervention for aortic valve dysfunction. | 1 month post procedure
  Composite measure of all-cause death, any stroke, VARC-3 type 1 (only overt bleeding that requires a transfusion of 1 unit of whole blood/red blood cells (BARC 3a), type 2 and 3 bleeding, AKI stage 2-4, rehospitalization for a procedure-related event or reintervention for aortic valve dysfunction.
Primary efficacy endpoint at 1 year (non-inferiority): Composite measure of all-cause death, any stroke, or rehospitalization for valve related event | 1 year post procedure
  Composite measure of all-cause death, any stroke, or rehospitalization for valve related event at 1 year (VARC-3 definition)
CT Scan Sub Study endpoints: primary endpoint : prevalence of feasible redoTAVR or ViV TAVR without requiring leaflet modifications techniques (green cases). | 1 month post procedure
  Proportion of participants classified as "green cases" (redo-TAVR or ViV-TAVR feasible without leaflet modification) based on predefined CT scan criteria, including annular dimensions, coronary access, and valve frame interactions.

SECONDARY OUTCOMES:
Secondary Endpoint: Individual components of the primary endpoints: all cause mortality over time | 1, 2, 3 and 5 years
  Number of participants who experience all-cause mortality at each follow-up time point.
Secondary Endpoint: Individual components of the primary endpoints: Stroke Over Time | 1, 2, 3 and 5 years
  Number of participants with any stroke (ischemic or hemorrhagic) as defined by clinical assessment and imaging confirmation.
Secondary Endpoint: Individual components of the primary endpoints: Bleeding Events (VARC-3 Type 1, 2, and 3) Over Time | 1, 2, 3 and 5 years
  Number of participants experiencing bleeding events classified as VARC-3 type 1 (BARC 3a), type 2 and 3.
  * Scoring System: Valve Academic Research Consortium (VARC) scale:
  * 1
    * Overt bleeding not requiringing surgical or percutaneous intervention, but requiring medical intervention, leading to hospitalization, an increased level of care, or medical evaluation
    * Overt bleeding requiring a transfusion of 1 unit of whole blood/RBC
  * 3
    * Overt bleeding in a critical organ, such as intracranial, intraspinal, intraocular, pericardial or intramuscular with compartment syndrome
    * Overt bleeding causing hypovolemic shock or severe hypotension
    * Overt bleeding requiring reoperation, surgical exploration, or re-intervention for the purpose of controlling bleeding
    * Post-thoracotomy chest tube output ≥2 L within 24-h
    * Overt bleeding requiring a transfusion of ≥5 units of whole blood/RBC
    * Overt bleeding associated with a haemoglobin drop ≥5 g/dL
  * Higher scores indicate worst outcomes
Secondary Endpoint: Individual components of the primary endpoints: Acute Kidney Injury (AKI) Stage 2-4 Over Time | 1, 2, 3 and 5 years
  Number of participants with acute kidney injury (AKI) stage 2-4 based on VARC-3
  * Scale Information: AKI from Valve Academic Research Consortium 3 (VARC-3):
    * Scoring System:
    * Stage 1: AKI that fulfils at least one of the following criteria:
  * Increase in serum creatinine ≥150-200% (≥1.5-2.0x increase) within 7 days compared with baseline
  * Increase of ≥ 0.3mg/dL (≥26.4 μmol/L) within 48 h of the index procedure
    o Stage 2: AKI that fulfils the following criterion:
  * Increase in serum creatinine >200-300% (>2.0-3.0x increase) within 7 days compared with baseline
    o Stage 3: AKI that fulfils at least one of the following criteria:
  * Increase in serum creatinine >300% (>3.0x increase) within 7 days compared with baseline
  * Serum creatinine ≥4.0 mg/dL (≥354 μmol/L) with an acute increase of ≥0.5 mg/dL (≥44 μmol/L)
    * Stage 4: AKI requiring new temporary or permanent renal replacement therapy
    * Interpretation: Higher stages indicate more severe kidney injury
Secondary Endpoint: Individual components of the primary endpoints: Rehospitalization for Procedure-Related Event Over Time | 1, 2, 3 and 5 years
  Number of participants requiring rehospitalization due to procedure-related complications.
Secondary Endpoint: Individual components of the primary endpoints: Reintervention for Aortic Valve Dysfunction Over Time | 1, 2, 3 and 5 years
  Number of participants requiring reintervention (redo-TAVR, SAVR, or valve explantation) due to aortic valve dysfunction.
Secondary Endpoint: Feasibility of re-TAVR based on CT scan evaluation (CT scan, for selected sites only) | 1 month post procedure
  Number of participants in whom redo-TAVR is deemed feasible based on CT scan evaluation.
  Feasibility will be assessed using predefined anatomical criteria, including:
  Annular dimensions Coronary access Valve frame interactions Need for leaflet modification techniques Feasibility will be categorized as: "Feasible without modification," "Feasible with modification," or "Not feasible.
Secondary Endpoint: Number of Participants Requiring New Permanent Pacemaker Implantation (PPI) Due to Conduction System Disturbances | 1 month post procedure
  Number of participants who require a new permanent pacemaker implantation (PPI) within 1 month post-procedure due to conduction system disturbances (e.g., high-degree atrioventricular block, left bundle branch block).
  Indications for PPI will be based on standard clinical guidelines.
Secondary Endpoint: Rate of prosthetic valve regurgitation (moderate or severe) | 1 year post procedure
Secondary Endpoint: Number of Participants with Major Vascular Complications (VARC-3 Criteria) | 1 month post procedure
  Number of participants experiencing major vascular complications within 1 month post-procedure, as defined by VARC-3 criteria.
  o Scoring System: Valve Academic Research Consortium-3 (VARC-3) criteria o Definition: MAJOR vacular complication: One of the following:
  • Aortic dissection or aortic rupture • Vascular injury or compartment syndrome resulting in death,VARC type ≥2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment • Distal embolization (non-cerebral) from a vascular source resulting in death, amputation, limb or visceral ischaemia, or irreversible end-organ damage • Unplanned endovascular or surgical intervention resulting in death, VARC type ≥2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment • Closure device failure resulting in death, VARC type ≥2 bleeding, limb or visceral ischaemia, or irreversible neurologic impairment
Secondary Endpoint: Performance of the aortic valve : Gradients (mean/max) assessed by TTE | 1 year and 3 years post procedure
  Mean and peak aortic valve gradients (mmHg) will be measured by transthoracic echocardiography (TTE) at each follow-up time point.
  Values will be reported as mean ± standard deviation (SD).
Secondary Endpoint: Performance of the aortic valve : paravalvular leakage (PVL) grade evaluated by transthoracic echocardiogram (TTE) | 1 year and 3 years post procedure
  Number of participants stratified by paravalvular leakage (PVL) grade (None, Mild, Moderate, Severe), as assessed by TTE.
  PVL severity will be determined based on echocardiographic parameters defined by the VARC-3 criteria.
Secondary Endpoint: Performance of the aortic valve : effective orifice are (EOA) evaluated by transthoracic echocardiogram (TTE) | 1 year and 3 years post procedure
  Effective orifice area (EOA) (cm²) measured using the continuity equation on TTE.
  Values will be reported as mean ± standard deviation (SD).
Secondary Endpoint: Number of Participants with Structural Valve Deterioration (VARC-3) and/or Requiring Redo-TAVR or Valve Explantation | 5 years post procedure
  Number of participants experiencing significant structural valve deterioration (SVD) as defined by VARC-3 criteria.
  SVD will be assessed by transthoracic echocardiography (TTE) Number of participants requiring redo-TAVR or surgical valve explantation within 5 years post-procedure.
CT Scan Sub Study endpoints: Secondary outcomes : feasibility of redoTAVR or ViV TAVR with or without requiring leaflet modification techniques | 1 month post procedure
  Proportion of participants in whom redo-TAVR or ViV-TAVR is feasible, with or without requiring leaflet modification techniques, based on CT scan evaluation. Classification will be based on predefined anatomic and hemodynamic feasibility criteria.
CT Scan Sub Study endpoints: Secondary outcomes: prevalence of HALT in both TAVR and SAVR groups | 1 month post procedure
  Number of participants with HALT detected on CT scan in both TAVR and SAVR groups. HALT will be defined as the presence of hypo-attenuated leaflet thickening observed on post-procedure CT imaging.
CT Scan Sub Study endpoints: Secondary outcomes: Impact of HALT on Mean Transvalvular Gradient - Valve Hemodynamics | 1 month post procedure
  * Outcome Measure: Mean change in mean transvalvular gradient (mmHg) in participants with and without HALT, measured by transthoracic echocardiography (TTE).
  * Time Frame: 1 month post-procedure
  * Unit of Measure: mmHg
  * Interpretation: A higher mean transvalvular gradient suggests increased valve obstruction.
CT Scan Sub Study endpoints: Secondary outcomes: Impact of HALT on Peak Transvalvular Gradient - Valve Hemodynamics | 1 month post procedure
  * Outcome Measure: Mean change in peak transvalvular gradient (mmHg) in participants with and without HALT, measured by transthoracic echocardiography (TTE).
  * Time Frame: 1 month post-procedure
  * Unit of Measure: mmHg
  * Interpretation: A higher peak transvalvular gradient indicates greater hemodynamic burden on the valve.
CT Scan Sub Study endpoints: Secondary outcomes: Impact of HALT on Effective Orifice Area (EOA) - Valve Hemodynamics | 1 month post procedure
  * Outcome Measure: Mean change in effective orifice area (cm²) in participants with and without HALT, measured by transthoracic echocardiography (TTE).
  * Time Frame: 1 month post-procedure
  * Unit of Measure: cm²
  * Interpretation: A lower EOA suggests impaired valve opening and increased risk of stenosis.
CT Scan Sub Study endpoints: Secondary outcomes: Mean Transvalvular Gradient - THV Hemodynamics | 1 month post procedure
  * Outcome Measure: Mean transvalvular gradient (mmHg) measured by TTE post-implantation.
  * Time Frame: 1 month post-procedure
  * Unit of Measure: mmHg
  * Interpretation: Higher gradients indicate increased obstruction.
CT Scan Sub Study endpoints: Secondary outcomes: Peak Transvalvular Gradient - THV Hemodynamics | 1 month post procedure
  * Outcome Measure: Peak transvalvular gradient (mmHg) measured by TTE post-implantation.
  * Time Frame: 1 month post-procedure
  * Unit of Measure: mmHg
  * Interpretation: Higher peaks indicate more severe stenosis.
CT Scan Sub Study endpoints: Secondary outcomes: Effective Orifice Area (EOA) - THV Hemodynamics | 1 month post procedure
  * Outcome Measure: Effective orifice area (cm²) measured by TTE post-implantation.
  * Time Frame: 1 month post-procedure
  * Unit of Measure: cm²
CT Scan Sub Study endpoints: Secondary outcomes: Commissural Alignment of THV | 1 month post procedure
  Mean commissural misalignment angle (degrees) measured by CT scan to evaluate THV positioning relative to native aortic valve commissures.

CONTACTS AND LOCATIONS:
Locations (7):
- France (5):
  - CHU Lille, Lille
  - Infirmerie Protestante de Lyon, Lyon
  - Massy-Hôpital Jacques Cartier, Massy
  - CHU de Rouen, Rouen
  - Clinique Pasteur, Toulouse
- Hospital clínico universitario de Valladolid, Valladolid, Spain
- CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Milojevic M, Myers PO, Falk V, Bavaria JE, Borger MA, Casselman FPA, Badhwar V, Kaul S, Siepe M, Sadaba JR. Methodological Appraisal of Ongoing Trial of Transcatheter Aortic Valve Implantation Versus Surgical Aortic Valve Replacement in Younger Patients: From Incentives to Guideline-Informing Evidence. Eur J Cardiothorac Surg. 2025 Dec 1;67(12):ezaf348. doi: 10.1093/ejcts/ezaf348. PMID 41351226